CLINICAL TRIAL: NCT02009436
Title: Phase I Study of Inhaled Vidaza® in Patients With Advanced NSCLC
Brief Title: Azacitidine in Treating Patients With Stage IV or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-382; NCI-2014-01269 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-382 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2013-10-21; First posted 2013-12-12 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine) (Experimental): Patients receive azacitidine via nebulizer over 20 minutes QD on days 1-5 and 15-19. Treatment repeats every 28 days for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients may continue treatment on a case-by-case basis at the discretion of principal investigator and Institutional Review Board.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Azacitidine — Given via nebulizer
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This pilot phase I trial studies the side effects and best dose of azacitidine in treating patients with lung cancer that is stage IV or has returned after previous treatments (recurrent). Azacitidine is a drug used in chemotherapy that may stop tumor cells from growing or spreading by activating genes that help prevent cancer growth, called tumor suppressor genes. As people age, these genes are silenced by a chemical reaction that occurs naturally in the body, or by exposure to environmental factors such as smoking. Azacitidine may help reverse this process and restore the function of the tumor suppressor genes. Delivering azacitidine directly into the lungs by inhalation may work better in treating lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and toxicity of inhaled Vidaza® (azacitidine) with special emphasis on pulmonary toxicity.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of inhaled Vidaza®. II. To determine the changes in global methylation patterns in the bronchial epithelium (bronchial tissue samples) pre and post treatment.

III. To determine the changes in methylation patterns in the exhaled breath. IV. To evaluate the efficacy of inhaled Vidaza® on intra-thoracic tumors (response rate by Response Evaluation Criteria in Solid Tumors [RECIST] criteria for intrapulmonary lesions).

V. To estimate the progression free, intra-thoracic tumor progression free and overall survival.

VI. To determine the minimum effective dose of inhaled Vidaza® required to induce changes in the methylation status and re-expression of a panel of genes, including 5 candidate tumor suppressor genes (cyclin-dependent kinase inhibitor 2A [p16], h-cadherin [H-Cad], opioid binding protein/cell adhesion molecule-like [OPCML], secreted frizzled-related protein 1 [SFRP-1], and ras association domain family 1 [RASSF1A]) that are silenced in 20-50% of bronchial tissue of heavy smokers with lung cancer.

OUTLINE: This is a dose-escalation study.

Patients receive azacitidine via nebulizer over 20 minutes once daily (QD) on days 1-5 and 15-19. Treatment repeats every 28 days for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients may continue treatment on a case-by-case basis at the discretion of principal investigator and Institutional Review Board.

After completion of study treatment, patients are followed up at 4-6 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of stage IV or recurrent non-small cell lung cancer (according to American Joint Committee on Cancer [AJCC] staging, 7th edition)
* Patient has received at least one prior standard chemotherapy or targeted therapy for treatment of lung cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) >= 1,500 cells/ul
* Platelets >= 100,000 cells/ul
* Hemoglobin >= 9.0 g/dl (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= g/dl is acceptable)
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin < 2.0 times the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x the ULN
* Adequate pulmonary reserve defined as adequate airflow defined by a measured forced expiratory volume (FEV1) not less than 50% of the predicted value and adequate pulmonary reserve as evidenced by a FEV1/forced vital capacity (FVC) ratio of 65% or greater
* Patient must sign study specific informed consent prior to study entry
* Women of childbearing potential must have:

  * A negative serum or urine pregnancy test (sensitivity =< 25 IU human chorionic gonadotropin [HCG]/L) within 72 hours prior to the start of study drug administration
  * Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy

Exclusion Criteria:

* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study
* Contraindication to or unwillingness to undergo study related procedures including a repeat bronchoscopy
* Participation in an investigational drug or device study or treatment with any antineoplastic agent within 14 days of the first day of dosing on this study
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* History of hypersensitivity to mannitol
* Unwillingness or inability to comply with the study protocol for any other reason
* Women who:

  * Are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
  * Have a positive pregnancy test at baseline, or
  * Are pregnant or breastfeeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Minimum effective dose of inhaled azacitidine, defined as the dose required to induce the re-expression of any of the relevant 5 candidate tumor suppressor genes by two fold between pre and post treatment bronchial biopsies in 50% of evaluable patients | Up to day 28 after the first course of treatment
  The data will be analyzed and presented in descriptive fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Perez-Soler, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Cheng H, Zou Y, Shah CD, Fan N, Bhagat TD, Gucalp R, Kim M, Verma A, Piperdi B, Spivack SD, Halmos B, Perez-Soler R. First-in-human study of inhaled Azacitidine in patients with advanced non-small cell lung cancer. Lung Cancer. 2021 Apr;154:99-104. doi: 10.1016/j.lungcan.2021.02.015. Epub 2021 Feb 17. PMID 33636454